CLINICAL TRIAL: NCT06371157
Title: A Phase III, Randomized, Double-blinded, Multicenter Study of Cadonilimab (AK104) + Lenvatinib in Combination With Transarterial Chemoembolization (TACE) Versus TACE in Participants With Incurable/Non-metastatic Hepatocellular Carcinoma
Brief Title: A Study of AK104+Lenvatinib in Combination With Transarterial Chemoembolization (TACE) Versus TACE in Participants With Incurable/Non-metastatic Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK104-308
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): AK104+ Lenvatinib in Combination With Transarterial Chemoembolization (TACE)
  Interventions: Drug: AK104; Drug: Lenvatinib; Procedure: TACE
- Arm B (Placebo Comparator): Placebo for AK104 + Placebo for Lenvatinib in Combination With TACE
  Interventions: Procedure: TACE; Other: Placebo for AK104; Other: Placebo for Lenvatinib
- Arm C (Other): AK104 + Placebo for Lenvatinib in Combination With TACE
  Interventions: Drug: AK104; Procedure: TACE; Other: Placebo for Lenvatinib

INTERVENTIONS:
Drug: AK104 — intravenous
  Arms: Arm A; Arm C
Drug: Lenvatinib — oral
  Arms: Arm A
Procedure: TACE — TACE (chemo and embolic agent injection into the hepatic artery)
Other: Placebo for AK104 — intravenous
  Arms: Arm B
Other: Placebo for Lenvatinib — oral
  Arms: Arm B; Arm C

SUMMARY:
A study to evaluate cadonilimab (AK104) + lenvatinib in combination with transarterial chemoembolization (TACE) versus TACE in participants with incurable/non-metastatic hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by histology/cytology，or meet the clinical diagnostic criteria of the American Association for the Study of Liver Diseases (AASLD)
2. No evidence of metastasis
3. Not amenable to curative surgery or transplantation or curative ablation but amenable to TACE
4. Child Pugh score class A
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
6. Measurable disease by RECIST 1.1
7. Adequate organ function

Exclusion Criteria:

1. History of liver transplantation
2. History of hepatic encephalopathy
3. Uncontrolled arterial hypertension
4. Deep venous thrombosis within 3 months before first treatment
5. Bleeding events within the last 6 months
6. Co-infection with HBV and HCV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented progressive disease or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1 as assessed by blinded independent central review (BICR).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 2 years
  OS is defined as the time from randomization to death due to any cause.
PFS per RECIST 1.1 | Up to approximately 2 years
  Assessed by investigators
Objective Response Rate (ORR) per RECIST 1.1 and Modified Response Evaluation Criteria in Solid Tumors (mRECIST) | Up to approximately 2 years
  Assessed by BICR and investigators
Duration of Response (DOR) per RECIST 1.1 and mRECIST | Up to approximately 2 years
  Assessed by BICR and investigators
Disease Control Rate (DCR) per RECIST 1.1 and mRECIST | Up to approximately 2 years
  Assessed by BICR and investigators
Time to Response (TTR) per RECIST 1.1 and mRECIST | Up to approximately 2 years
  Assessed by BICR and investigators

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Shao, MD, Principal Investigator — Zhejiang Cancer Hospital; Gaojun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (4):
- China (4):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang